CLINICAL TRIAL: NCT01850225
Title: A Feasibility Study of the Placement, Use, and Safety of the Nucleus 24 Auditory Brainstem Implant in Non-Neurofibromatosis Type 2 (NF2) Pediatric Patients
Brief Title: Feasibility Study of Auditory Brainstem Implant in Young Children
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: House Research Institute (Other)
Collaborators: House Clinic, Inc. (Industry); Children's Hospital Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ped ABI
Record Dates: First submitted 2013-04-24; First posted 2013-05-09 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2013-10

CONDITIONS: Bilateral Cochlear Aplasia; Bilateral Cochlear Nerve Deficiency; Bilateral Cochlear Ossification Secondary to Meningitis
MeSH Terms: interventions — Auditory Brain Stem Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device implantation (Experimental): Implantation of device
  Interventions: Device: Auditory brainstem implant

INTERVENTIONS:
Device: Auditory brainstem implant
  Other Names: Cochlear Corporation Nucleus 24

SUMMARY:
Current treatment options for bilateral profoundly deaf children, diagnosed with inner ear anatomical abnormalities are limited, and in the case of absent cochleas, non-existent. An auditory brainstem implant (ABI) places an electrode close to the auditory nucleus in the brainstem. Children aged 2 - 5 who are not candidates for a cochlear implant, or who did not demonstrate benefit from a cochlear implant, will be implanted with an ABI and followed for 1 year for safety and a total of 3 years for preliminary efficacy. This is a feasibility study to determine the safety of the ABI.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral profound deafness due to cochlear aplasia, cochlear nerve deficiency, or ossification secondary to meningitis
* If previously received a cochlear implant, must demonstrate lack of benefit from that device

Exclusion Criteria:

* Medical contraindication to craniotomy/intracranial surgery
* Severe cognitive or developmental delays

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Number of Serious Adverse Events | 12-month post-activation
  Count of the number of expected serious adverse events must not exceed that known to occur in pediatric retrosigmoid craniotomy and Count of the number of unexpected serious adverse events must not exceed 2 in the first 5 children.

SECONDARY OUTCOMES:
Access to sound at a level (dB) and within the frequency range (500-4000 Hz), known to be associated with speech | 3 years post-activation
  ability to detect sounds

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wilkinson, MD, Principal Investigator — House Research Institute; Laurie Eisenberg, PhD, Principal Investigator — House Research Institute
Locations (1):
- House Research Institute CARE Center, Los Angeles, California, United States